CLINICAL TRIAL: NCT04957433
Title: Lung Health Check Biomarker Study
Brief Title: 'Lung Health Check' Biomarker Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Imperial College London (Other); Royal Marsden Partners Cancer Alliance (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCR5067
Record Dates: First submitted 2020-01-13; First posted 2021-07-12 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Lung Cancer; Cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort A: Patients new to The Lung Health Check (TLHC) pilot who are attending their first lung health check
  Interventions: Diagnostic Test: Blood Specimen
- Cohort B (Nodule Suveillance): Patients who have already undergone one lung health check as part of the TLHC programme, and are now being followed up at 3 months (B1), 12 months (B2) or other (BX) due to an indeterminate finding (e.g. lung nodule)
  Interventions: Diagnostic Test: Blood Specimen
- Cohort C (Incident Scan): Patients who are already part of TLHC attending for routine 'incident' round follow-up scanning (usually at approximately 24 months)
  Interventions: Diagnostic Test: Blood Specimen
- Cohort D: Participants with interstitial lung abnormalities (ILAs) identified as part of TLHC, who are referred to the interstitial lung disease (ILD) unit at Royal Brompton Hospital.
  Interventions: Diagnostic Test: Blood Specimen

INTERVENTIONS:
Diagnostic Test: Blood Specimen — Blood and Sputum Specimen Samples
  Other Names: Sputum Specimen

SUMMARY:
CT screening of lung cancer offers an opportunity to diagnose early stage lung cancers which is associated with better prognosis - indeterminate results delay diagnosis whilst interval imaging is awaited to assess risk of cancer. This study will allow us to examine the potential of blood-based biomarkers to augment CT screening for lung cancer.

Hypotheses

1. Blood and sputum samples can be collected in patients attending lung health checks as part of the Lung Health Check pilot in West London at fixed and mobile scanners and safely transported for processing and storage in preparation for biomarker development.
2. The biomarkers will help to identify cohorts of

   1. High-risk patients in whom CT surveillance should be conducted more readily/frequently and diagnostic procedures performed earlier.
   2. Low-risk patients who might need reduced surveillance intensity.
   3. Patients with interstitial lung abnormalities that share similar biomarker characteristics to patients with clinically significant interstitial lung disease

DETAILED DESCRIPTION:
1. Background 1.1 Lung cancer & CT screening Over 46,000 cases of lung cancer are diagnosed every year in the UK, making it the 3rd most common cancer type. Lung cancer is the biggest cause of cancer mortality in the UK and worldwide due to late presentation in the majority of cases. One year survival for lung cancer ranges from 83% at stage I to 17% in stage IV disease (CRUK data).

   Reduced lung cancer mortality (20-26%) can be achieved by Lung Health Checks - which use 'low dose' CT (LDCT) scans of high-risk populations (e.g. heavy smokers), by increasing the proportion of cases diagnosed at an earlier stage when the treatment options are better (National Lung Cancer Screening Trial and NELSON studies). A number of pilot trials within the UK have led to a commitment by NHS England to roll-out a £70m national pilot. RM Partners commenced recruitment to one of the earlier pilots across two clinical commissioning groups (CCGs) in West London in 2018, inviting approximately 1000 patients for an LDCT scan at a fixed and mobile scanner (based in a supermarket car park). This pilot will be extended in 2019-2020 with a further 1000-2000 patients - this will include both new patients and others who will have a 24 month 'incident scan' to re-examine for any new cancer after a previously normal baseline scan). This study will test the uptake and feasibility of biomarker testing and potential scientific opportunities from specimens received.

   1.2 Current Limitations of Lung Health Checks A) Patient Selection: Two lung cancer risk calculators, the modified Liverpool Lung Project (LLPv2) and the Prostate, Lung, Colorectal and Ovarian Cancer Screening Trial (PLCO) are both multivariate risk prediction models which have been used to select patients for screening. Both models have been used to support the identification of high risk individuals during the Lung Health Check pilot to determine the risk of lung cancer and stratifying for LDCT screens. Improved patient selection has been identified as a priority to improve the sensitivity and specificity of lung health checks.

   B) Indeterminate Findings: In addition management of indeterminate 'nodules' which can be either small, possibly early cancers, or benign scarring requires delayed e.g. 3 or 12 month surveillance scans to stratify more invasive procedures such as lung biopsy to confirm the diagnosis. Blood biomarkers capable of identifying patients at increased risk of developing or harbouring lung cancer would be valuable adjuncts to protocols for surveillance and invasive monitoring. Nodules are seen in approximately 10% of scans.

   Existing clinical scores (e.g. Brock score) could be improved upon (see British Thoracic Society guidelines) and there remains significant clinical uncertainty about best management in patients with indeterminate nodules.

   1.3 Circulating and sputum biomarkers in lung cancer early diagnosis Identification of blood-based biomarkers is an important priority of lung health check research. Integrating biomarker data along with nodule size and/or volume with other radiological indices may enable improved risk stratification of surveillance, identifying those at high risk of lung cancer and requiring more frequent following up, versus those at low risk and requiring less follow up.

   Current technology recognises the potential to detect tumour specific proteins, metabolites or cell free DNA are examples of biological material in the circulating blood of patients with lung cancer. Existing approaches under investigation include genomics, epigenomics, microbiomics, gene methylation and metabolomics. Some groups have also looked at circulating tumour cells and immune responses to identify patients with higher risk of cancer. There is also a growing interest in using other bodily fluids, such as sputum, for this purpose. These have not reached readiness for clinical studies thus far but in other tumour types, such as in bowel cancer equivalent tests such as the nationally commissioned stool biomarker ('FIT test) improve diagnostic yield of bowel cancer screening to stratify resources more cost-effectively.

   Existing approaches in lung cancer screening research suggests that further work will be needed to identify circulating DNA from the smallest lesions where sensitivity remains highly variable between studies (10-100%) depending upon the technique selected and the stage of disease. There is a continued need to explore the role of these approaches in lung cancer early diagnosis populations, which will likely require a multi-modality approach of several technologies, for example combining genomics imaging biomarkers with radiomics. Sputum sensitivity has been shown previously to be in excess of 50% in a number of settings
2. Rationale CT screening of lung cancer offers the opportunity to diagnose early stage lung cancers which is associated with better prognosis - indeterminate results delay diagnosis whilst interval imaging is awaited to assess risk of cancer. This study will allow the investigators to examine the potential of blood-based biomarkers to augment CT screening for lung cancer.

Poor patient uptake and logistical issues are perceived to be key challenges to CT screening that may preclude clinical utility of a blood/sputum biomarker. Assessing whether such biomarkers can contribute to clinical decision making could then be explored.

Technologies for choosing laboratory biomarkers for risk stratification is evolving rapidly. Currently there is interest in genomics and circulating tumour cells, but as the potential for epigenomics, metabolomics, proteomics and exosome analysis evolve, the investigators hope to have prepared a suitable biobank with which can be used to challenge the latest of these approaches to the aim of stratification. This may be derived from germline or tumour-based markers of risk or be derived from the interaction between the tumour cells, host and immune response.

3. Hypothesis

1. Blood and sputum samples can be collected in patients attending lung health checks as part of the Lung Health Check pilot in West London at fixed and mobile scanners and safely transported for processing and storage in preparation for biomarker development.
2. The biomarkers will help to identify cohorts of

   1. High-risk patients in whom CT surveillance should be conducted more readily/frequently and diagnostic procedures performed earlier.
   2. Low-risk patients who might need reduced surveillance intensity.

7. Methodology This study is designed to collect sputum and blood specimens for laboratory development of a biomarker that will guide stratification and personalisation of CT screening study interval. The investigators seek access to basic, link-anonymized clinical and imaging data which can be integrated with data obtained from the sputum/blood biomarkers - this will be linked by the study ID number.

These data are not expected to influence clinical decision-making. There are no routine clinical arrangements in place to account for research findings. If a result is identified for which there is concern, which could be significant for the patient's care, the principle investigator will seek advice from the patient's clinical team. This is discussed in the patient information sheet and consent form.

This is a collaborative research project across RM Partners, Royal Brompton & Harefield Hospitals NHS Foundation Trust, Royal Marsden Hospital NHS Foundation Trust, and Imperial College London.

ELIGIBILITY:
Inclusion Criteria:

* Patients invited to participate in the Royal Marsden (RM) Partners Lung Health Check pilot study who undergo one or more CT scans:
* Between the age of 55-75 years of age; and
* Current smokers or ex-smokers who have quit after the age of 40.

Exclusion Criteria:

* Patients excluded from the Lung Health Check:
* On the palliative care register;
* Any active malignancy undergoing treatment
* Daily activity levels equivalent to performance score 3 or 4; and
* Unable to consent to Lung Health Check Biomarker Study

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had been identified using two lung cancer risk calculators, the modified Liverpool Lung Project (LLPv2) and the Prostate, Lung, Colorectal and Ovarian Cancer Screening Trial (PLCO) to be at high risk for lung cancer and recruited to The Lung Health Check (TLHC) pilot taking place in West London.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the primary objective to collate a lung health check biobank | 2 Years
  The feasibility of the primary objective to collate a lung health check biobank will be reported as a percentage after the final participant recruited has donated both a baseline sample and also their final specimen (or on the same date should they decline to do so). The primary end point of the project will be considered feasible if consent to a blood test, collection and storage can be achieved in at least 50% of the 1000 patients approached for the biomarker study who undertake an LDCT scan.

SECONDARY OUTCOMES:
Confirming if a lung cancer genomics panel differs between participants who receive a diagnosis of lung cancer at the time of the baseline scan and those who do not | 2 Years
  The first secondary end point will be met if, a lung cancer genomics panel on sputum/peripheral blood samples taken at the time of the baseline LDCT screening scans differs between participants who receive a diagnosis of lung cancer at the time of the baseline scan (or associated biopsy) and those whom do not.
Confirming if a lung cancer genomics panel (taken at baseline LDCT screening scans) differs between those who receive a diagnosis of lung cancer and those who do not after completion of follow-up imaging | 2 years
  An additional secondary end point will be met if a lung cancer genomics panel on sputum or peripheral blood samples taken at baseline LDCT screening scans differs between patients who receive a diagnosis of lung cancer after completion of follow-up imaging (or two years, whichever occurs sooner) and those whom do not.
Confirming if peripheral blood telomere length can determine those who have interstitial lung abnormalities at those who do not, and who is at higher risk of developing overt pulmonary fibrosis | 2 years
  An additional secondary endpoint will be met if peripheral blood telomere length differs between those with interstitial lung abnormality and without and can predict those at higher risk of developing overt pulmonary fibrosis

OTHER OUTCOMES:
Are sputum and blood specimens of suitable volume and quality for given proposed laboratory biomarker tests | 2 Years
  The exploratory endpoints are indicators of whether for a given proposed laboratory biomarker test the sputum and blood specimens are deemed of suitable volume/quality to be subjected to the given laboratory approach (e.g. in the case of genomic analysis, this could be quantified as sample volume and DNA content RIN (RNA integrity number) as will be dictated by the laboratory protocol
Do given biomarker panels differ between patients who receive a diagnosis of lung cancer and those who do not. | 2 years
  The exploratory endpoints are indicators of whether for a given proposed laboratory biomarker test A given biomarker panel on sputum and/or peripheral blood samples and/or histopathological analysis of routine specimens (±combined clinical or imaging data) taken at the time of baseline LDCT screening scans differs between patients who receive a diagnosis of lung cancer after completion of follow-up imaging (or two years, whichever occurs sooner) and those whom do not.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Brompton NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cohen JD, Li L, Wang Y, Thoburn C, Afsari B, Danilova L, Douville C, Javed AA, Wong F, Mattox A, Hruban RH, Wolfgang CL, Goggins MG, Dal Molin M, Wang TL, Roden R, Klein AP, Ptak J, Dobbyn L, Schaefer J, Silliman N, Popoli M, Vogelstein JT, Browne JD, Schoen RE, Brand RE, Tie J, Gibbs P, Wong HL, Mansfield AS, Jen J, Hanash SM, Falconi M, Allen PJ, Zhou S, Bettegowda C, Diaz LA Jr, Tomasetti C, Kinzler KW, Vogelstein B, Lennon AM, Papadopoulos N. Detection and localization of surgically resectable cancers with a multi-analyte blood test. Science. 2018 Feb 23;359(6378):926-930. doi: 10.1126/science.aar3247. Epub 2018 Jan 18. PMID 29348365
- [Result] Wang BH, Li YY, Han JZ, Zhou LY, Lv YQ, Zhang HL, Zhao L. Gene methylation as a powerful biomarker for detection and screening of non-small cell lung cancer in blood. Oncotarget. 2017 May 9;8(19):31692-31704. doi: 10.18632/oncotarget.15919. PMID 28404957
- [Result] Newman AM, Bratman SV, To J, Wynne JF, Eclov NC, Modlin LA, Liu CL, Neal JW, Wakelee HA, Merritt RE, Shrager JB, Loo BW Jr, Alizadeh AA, Diehn M. An ultrasensitive method for quantitating circulating tumor DNA with broad patient coverage. Nat Med. 2014 May;20(5):548-54. doi: 10.1038/nm.3519. Epub 2014 Apr 6. PMID 24705333
- [Result] Ye M, Li S, Huang W, Wang C, Liu L, Liu J, Liu J, Pan H, Deng Q, Tang H, Jiang L, Huang W, Chen X, Shao D, Peng Z, Wu R, Zhong J, Wang Z, Zhang X, Kristiansen K, Wang J, Yin Y, Mao M, He J, Liang W. Comprehensive targeted super-deep next generation sequencing enhances differential diagnosis of solitary pulmonary nodules. J Thorac Dis. 2018 Apr;10(Suppl 7):S820-S829. doi: 10.21037/jtd.2018.04.09. PMID 29780628
- [Result] Zhao H, Chen KZ, Hui BG, Zhang K, Yang F, Wang J. Role of circulating tumor DNA in the management of early-stage lung cancer. Thorac Cancer. 2018 May;9(5):509-515. doi: 10.1111/1759-7714.12622. Epub 2018 Mar 12. PMID 29528556